CLINICAL TRIAL: NCT01866878
Title: Rehabilitation Protocol for Disorders on Hand Sensitivity in Multiple Sclerosis Patients.
Acronym: FINGER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-PP-13
Record Dates: First submitted 2013-04-30; First posted 2013-06-03 (Estimated); Last update posted 2025-12-02 (Actual); Status verified 2018-03

CONDITIONS: Multiple Sclerosis
Keywords: transcutaneous electrical nerve stimulation, sensitivity, multiple sclerosis,Reeducation through labor tactile discrimination
MeSH Terms: conditions — Multiple Sclerosis; Hypersensitivity | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A group enjoying a corrective touch (Experimental): At first, the patient is asked to gradually define the different types of touch that is applied to the hyposensitive area (fixed or mobile touches) with different textures and then compare them with the healthy side. In a second step, the patient is asked to associate multiple items sensation shape and texture, shape and weight. In a third step is used everyday objects.
  Desensitisation techniques find their interest mainly when symptoms or dysesthetic hyperesthésique. The objective is to increase the threshold of sensitivity to textures and particles eventually reduce dysaesthetic sensations.
  The patient class in order of increasing tolerance 10 textures. Dysesthetic area is stimulated 5 to 10 minutes by the first texture to numb the area by saturation of the action potential. This helps promote functional work and recognition of objects. As soon as the texture causes more trouble we go to the next texture by applying the same job.
  Interventions: Device: equipment rehabilitation stereognosis
- A group receiving TENS (TENS) (Experimental): Well known in the management of neuropathic pain based on the gate control theory, the application of TENS in the rehabilitation of touch remains to be demonstrated. A recent study applied to the September highlighted the long-term interest of the transcutaneous electrical nerve stimulation (TENS) to improve sensitivity tact arguing possible action on brain plasticity.
  Interventions: Device: TENS
- A control group (No Intervention)

INTERVENTIONS:
Device: equipment rehabilitation stereognosis
  Arms: A group enjoying a corrective touch
Device: TENS
  Arms: A group receiving TENS (TENS)

SUMMARY:
Sensory disorders in patients with multiple sclerosis are among the most common symptoms encountered.

A functional impairment based on sensory disorders of the hand. The hand is a sensory organ that transmits the cerebral cortex protopathic sensitive information, proprioceptive or epicritiques. The view-hand association plays an important role in the understanding of the environment. Its exploratory use remains an essential and voluntary basis. The process of recognition of the object passes through manipulation, but operates instantaneously. The brain is able to do a quick summary of the information it receives to determine the nature of the manipulated object. The exploration takes a posteriori, the brain can then determine the details component object (texture, shape, composition, temperature and weight).

Neurophysiological mechanisms that would explain the analgesic effects of transcutaneous electrical nerve stimulation (TENS) are not fully understood. Several theories underlying its use as a neuromodulator of pain. The gate control theory has led to the development of TENS devices. Recruitment of myelinated, large caliber, by the TENS electrodes afferent fibers increases the control exerted on spinal level, thereby inhibiting the action of afferent fibers of small caliber related to nociception. This stimulation strengthens the blocking of "gate" at the corresponding cell bodies of spinothalamic tract and reduces the transmission of nociceptive impulses to the spinal cord dorsal horn. This is segmental presynaptic inhibition depends on the area and stimulated.

The objective of this study is to improve the quality of life through improved sensitivity disorders of the hand in patients with MS, thanks to reeducation of the hand.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsing remitting MS defined according to Poser criteria [9] and McDonald [5].
* Age ≥ 18 years, male or female sex
* Patients with sensory disorders interesting hands, evidenced by clinical examination objective.
* Patients with an EDSS between 2 and 4 with functional sensitivity parameter ≥ 2.
* Patients affiliated to a social security scheme.
* Patients signed informed consent for the study.

Exclusion Criteria:

* Patients with other central or peripheral disorders may affect the sensitivity of the hand.
* Patients with allodynia in the study area
* Patients with a motor and / or deficit cerebellar ataxia of the upper limbs.
* Patients treated with psychotropic or antiepileptic drugs.
* Patients for whom a flare occurred affecting the sensitivity of the hand, within 30 days before enrollment.
* Patients holders of an active implantable medical device.
* Pregnant women and vulnerable patient population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-07-30 (Actual); Primary Completion 2015-07-28 (Actual); Study Completion 2015-07-28 (Actual)

PRIMARY OUTCOMES:
Compare quality of life between baseline and procedure | frist day, 1 month and 3 month
  Improve the quality of life through improved sensitivity disorders of the hand in patients with MS, thanks to reeducation of the hand.
  Unit of mesure: scale MusiQoL

SECONDARY OUTCOMES:
Compare the performance during functional tests between baseline and procedure | first day, 1 month and 3 month
  Improve performance of MS patients during functional tests in patients undergoing rehabilitation treatment compared to the control group.
  Using picking up test and thr Nine Hole Peg Test
Compare the improvement clinically sensitive target from baseline procedure | first day, 1 month and 3 month
  Improve clinically sensitive target of MS patients through a rehabilitation treatment compared to the control group.
  Using the Threshold pressure, the Threshold to the vibration and the Weber test.

CONTACTS AND LOCATIONS:
Overall Officials: Mikael COHEN, Medical Doctor, Study Director — Centre Hospitalier Universitaire de Nice
Locations (1):
- Hôpital Pasteur, Nice, France